CLINICAL TRIAL: NCT01909700
Title: Single Incision Pelvic Floor Mesh Implants
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011041
Record Dates: First submitted 2013-07-24; First posted 2013-07-26 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2013-07

CONDITIONS: Intra-operative Complications; Post Operative Complications
Keywords: Single Incision, Mesh, Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Incision Mesh (Experimental): intervention: single incision mesh implantation
  Interventions: Device: Single Incision Mesh

INTERVENTIONS:
Device: Single Incision Mesh — Single Incision Mesh is implanted for pelvic floor reconstruction

SUMMARY:
Objectives: To evaluate whether the use of single incision un-anchored small mesh implants is feasible, safe and effective for women with moderate pelvic organ prolapse.

Design: Patients diagnosed with moderate pelvic organ prolapse were enrolled to undergo a single incision un-anchored mesh operation. Follow-up was 4 to 23 months. The outcome measures for this study were the operative safety and post-operative pain, adverse effects and anatomical as well as functional cure.

Setting: The operations were performed under general anesthesia according with the reported surgical techniques at university and private hospitals.

DETAILED DESCRIPTION:
Eligibility criteria: female patients with moderate pelvic organ prolapse Outcome measures: intra operative safety and surgical complications, post operative complications and objective as well as subjective cure rates

ELIGIBILITY:
Inclusion Criteria:

* Patients with Gr 2-3 Pelvic Organ Prolapse

Exclusion Criteria:

*Previous Pelvic irradiation

Ages: 30 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2011-07; Primary Completion 2011-11 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Operative mesh related complications | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Menahem Neuman, Prof., Principal Investigator — Western Galilee MC Nahariya
Locations (1):
- Assuta MC, Tel Aviv, Israel